CLINICAL TRIAL: NCT05797805
Title: A Phase 1/2 Exploratory Study of the TBL1 Inhibitor, Tegavivint (BC2059), in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Tegavivint (BC2059) in Patients With Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iterion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITER-002-HCC
Record Dates: First submitted 2023-03-08; First posted 2023-04-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tegavivint single agent dosing regimen (Experimental): Tegavivint as monotherapy
  Interventions: Drug: Tegavivint
- Tegavivint plus cabozantinib combination dosing regimen (Experimental): Tegavivint in combination with cabozantinib
  Interventions: Drug: Tegavivint; Drug: Cabozantinib
- Tegavivint plus lenvatinib combination dosing regimen (Experimental): Tegavivint in combination with lenvatinib
  Interventions: Drug: Tegavivint; Drug: Lenvatinib

INTERVENTIONS:
Drug: Tegavivint — The first part is a phase 1 single-agent dose escalation, optimization, and expansion study of tegavivint in patients with advanced HCC after failure of at least one line of prior systemic therapy.
  Tegavivint single agent dosing regimen: Tegavivint will be administered weekly on Days 1, 8, 15, and 22 of a 28-day cycle
  Other Names: BC2059
Drug: Lenvatinib — In the second part of the study, the combination of tegavivint plus lenvatinib will be assessed with a limited dose escalation followed by a randomized dose optimization.
  Tegavivint plus lenvatinib combination dosing regimen: Tegavivint will be administered weekly on Days 1, 8, and 15 and 22 of a 28-day cycle; lenvatinib 8 mg (patients < 60 kg) or 12 mg (patients ≥ 60 kg) will be administered once daily on days 1-28 of a 28-day cycle .
  Other Names: Lenvima
  Arms: Tegavivint plus lenvatinib combination dosing regimen
Drug: Cabozantinib — In the second part of the study, the combination of tegavivint plus cabozantinib will be assessed with a limited dose escalation followed by a randomized dose optimization.
  Tegavivint plus cabozantinib combination dosing regimen: Tegavivint will be administered weekly on Days 1, 8, and 15 and 22 of a 28-day cycle; cabozantinib 60 mg (patients with Child-Pugh A) or 40 mg (patients with Child-Pugh B) will be administered orally once daily on days 1 through 28 of each 28-day cycle
  Other Names: cabometyx
  Arms: Tegavivint plus cabozantinib combination dosing regimen

SUMMARY:
This study will be conducted in 2 parts. The first part is a phase 1 single-agent dose escalation, and dose optimization, study of tegavivint in patients with advanced HCC after failure of at least one line of prior systemic therapy. The second part of the study will begin with a brief dose escalation part for each combination (tegavivint plus cabozantinib or tegavivint plus lenvatinib) followed by a combination dose expansion.

DETAILED DESCRIPTION:
This study will be conducted in patients with advanced hepatocellular carcinoma (HCC) who have progressed after at least one prior line of systemic therapy.

Tegavivint will be administered as a single agent first in a dose escalation and optimization design. Single agent dose escalation will follow a standard 3+3 design to determine the tegavivint maximum tolerated dose (MTD). Upon completion of the dose escalation design and review of all available safety, efficacy, PK and PD data the Safety Review Committee (SRC) will recommend two dose levels for dose selection optimization. The dose selection optimization will expand the two dose levels to approximately 20 patients randomized (1:1) per dose level (approximately 40 patients total) before declaring the recommended phase 2 dose (RP2D).

If sufficient clinical benefit is observed, the combination of tegavivint plus cabozantinib and tegavivint plus lenvatinib will be explored in the second part of the study. The second part of the study will begin with a brief dose escalation part for each combination (tegavivint plus cabozantinib or tegavivint plus lenvatinib). The starting dose level of tegavivint will be decided by the SRC and will start at either one dose level below the MTD or at a lower dose as defined by the SRC. The dose escalations will follow a standard 3+3 design, and the dose escalation increments for tegavivint will follow the monotherapy dose escalation schedule to determine the combinations MTDs. Upon completion of the combination dose escalations, approximately 12 additional patients will be enrolled in each combination arm at the tegavivint combination MTDs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Confirmed diagnosis of HCC by either:

Histologically or cytologically documented HCC based on pathology report or Clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria

* Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Child-Pugh class A or ≤ 7 class B liver score (no hepatic encephalopathy) within 7 days of first dose of the investigational product(s)
* Disease progression, intolerance or contraindication to at least one line of systemic therapy for advanced HCC Prior treatment with cabozantinib or lenvatinib is allowed in the combination dose escalation and expansion parts of the study.
* Measurable disease as defined by RECIST 1.1 with spiral computerized tomography (CT) scan or magnetic resonance imaging (MRI). Lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if progression has been demonstrated in such lesions.
* Willingness and ability to provide tumor biopsies during screening and while on treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to the first dose of the investigational product(s)
* Patients must have organ and marrow function as defined below within 7 days of the first dose of the investigational product(s):

  * Absolute neutrophil count (ANC) ≥ 1.2 x 109/L
  * Platelets ≥ 60 x 10^9/L; no transfusion within 7 days prior to assessment
  * Hemoglobin ≥ 9 g/dL (red blood cell transfusion or growth factors support is not allowed in the 14 days prior to the screening laboratory assessment)
  * Total bilirubin ≤ ULN
  * AST and ALT ≤ 5 x ULN
  * Renal Function : Estimated creatinine clearance (CrCl) ≥ 50 mL/min by the Cockcroft-Gault equation using actual body weight, or Estimated Glomerular Filtration Rate (eGFR) ≥ 50 mL/min/1.73m2 by CKD-EPI Creatinine Equation, or Measured creatinine clearance ≥ 50 mL/min
  * Albumin ≥ 2.8 g/dL
  * International normalized ratio (INR) ≤ 1.7, unless the patient is receiving anticoagulant therapy as long as the patient is within therapeutic range of intended use of anticoagulants
* Washout period prior to Day 1 of Cycle 1:

  * At least 21 days from the last dose of prior systemic anticancer treatment
  * At least 14 days from palliative radiotherapy (≤ 10 fractions or ≤30 gray [Gy] total dose or at least 28 days from radiotherapy > 30 Gy) to extrahepatic tumor lesions
  * At least 28 days from local or loco-regional therapy of intrahepatic tumor lesions (e.g. surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation)
* Grade ≤ 1 toxicity due to any previous cancer therapy according to the NCI-CTCAE, v.5. Grade 2 is allowed in case of alopecia and/or peripheral sensory neuropathy.
* Participants with past HCV infection will be eligible for the study. The treated participants must have completed their treatment at least 1 month prior to starting study intervention and HCV viral load must be below the limit of quantification.
* Participants with controlled HBV will be eligible if they meet the following criteria:

  * Antiviral therapy for HBV must be given for at least 4 weeks and HBV viral load must be less than 500 IU/mL prior to first dose of study drug. Patients on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study intervention.
  * Patients who are positive for anti-hepatitis B core antibody HBc, negative for hepatitis B surface antigen (HBsAg), and negative or positive for anti-hepatitis B surface antibody (HBs), and who have an HBV viral load under 100 IU/mL, do not require HBV antiviral prophylaxis.
  * Patients must have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤ 150/90 mm Hg at Screening and no change in antihypertensive medications within 1 week before Cycle 1 Day 1.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Patients receiving therapy with other anti-neoplastic or experimental agents
* Patients receiving concomitant strong inhibitors of CYP3A4/5 that cannot be discontinued 7 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* Patients receiving concomitant inducers of CYP3A4/5 that cannot be discontinued at least 14 days prior to Cycle 1 Day 1.
* Patients with known history of Gilbert's syndrome or other genetic conditions affecting UGT1A1 function.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tegavivint, or other agents used in study
* Malignant disease, other than that being treated in this study. Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) who have undergone potentially curative therapy are not excluded. Other exceptions include malignancies that were treated curatively and have not recurred within 3 years prior to Cycle 1 Day 1 and any malignancy considered indolent and that has never required therapy.
* Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
* Known central nervous system (CNS) involvement
* Uncontrolled concurrent illness including, but not limited to:

  * Ongoing or active infection (exception: HBV infection - see inclusion criteria)
  * Unhealed wounds or presence of any external drainage
  * Psychiatric illness/social situations that would limit compliance with study requirements; discuss with Medical Monitor if there are any questions
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  * Congestive heart failure, NYHA > Class II
  * Left ventricular ejection fraction < 50%
  * Unstable angina pectoris or cardiac arrhythmia
  * Baseline QTc (Fridericia) ≥ 450 milliseconds. In the event a QTc (Fridericia) measurement is not possible due to factors such as a pacemaker or bundle branch block, the patient may be evaluated by a cardiologist who must document no apparent increased risk for Torsades de Point or other morbidity associated with prolonged QTc. With such documentation, the patient may be eligible based with additional Medical Monitor review.
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
  * Myocardial infarct within 6 months before Cycle 1 Day 1
  * Clinically significant pericardial disease
* Any major surgery within 21 days prior to Cycle 1 Day 1. Major surgery is defined as any significantly invasive procedure into a major body cavity (abdomen, cranium etc.) and/or surgery requiring extensive recuperation (joint replacement). Please discuss with the Medical Monitor if there are any questions.
* Pregnant and breastfeeding women are excluded from this study. The effects of tegavivint on the developing human fetus have the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with tegavivint
* Women of child-bearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use one highly effective method of contraception, including hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device or intrauterine system; vasectomy or tubal ligation; and one effective method of contraception, including male condom, female condom, cervical cap, diaphragm or contraceptive sponge or abstaining from sex for the duration of study participation and for at least 4 months following completion of tegavivint and pembrolizumab (if applicable) administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with tegavivint.
* Exclusions for patients treated on study with cabozantinib or lenvatinib:

  * Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention: beta blockers or endoscopic treatment. Assessment of esophageal varices for patients in whom conventional medical intervention for known esophageal varices is already in place should be performed by endoscopy as per local standard of care.
  * Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management).
  * Persistent proteinuria of NCI-CTCAE version 5.0 grade 3 or higher. Urine dipstick result of 3+ is allowed if protein excretion (estimated by urine protein/creatinine ratio on a random urine sample) is <3.5 g/24 hours.
  * Clinically significant bleeding NCI-CTCAE version 5.0 grade ≥ 3 within 30 days before randomization.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months before the start of study medication.
  * Patients treated with medications with a known potential to prolong the QT/QTc interval.
  * Hypersensitivity or intolerance to cabozantinib (patients with hypersensitivity or intolerance to cabozantinib may enroll in treatment arms exploring tegavivint plus lenvatinib if they did not have hypersensitivity or intolerance to lenvatinib).
  * Hypersensitivity or intolerance to lenvatinib (patients with hypersensitivity or intolerance to lenvatinib may enroll in treatment arms exploring tegavivint plus cabozantinib if they did not have prior hypersensitivity or intolerance to cabozantinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | from the date of the first dose of study medication up to 90 days following last dose of study medication or initiation of new systemic anti-cancer therapy, whichever occurs first, an average of 1 year.
  Adverse events will be assessed according to the NCI-CTCAE version 5.0
Number of participants with dose limiting toxicities | Within a 28-day period after first dose of the study medication as a single agent or in combination with cabozantinib or lenvatinib.
  Dose limiting toxicities defined as a Grade 3 or greater adverse event as assessed by NCI-CTCAE version 5.0 (excluding toxicities clearly related to the underlying disease [HCC], disease progression, concomitant medications, or baseline concurrent medical conditions),and that meets any of the criteria included in Table 6-5.
Evaluate efficacy of tegavivint as a single agent | Tumors will be assessed at baseline and every 8 weeks until end of treatment, an average of 1 year
  Evaluate efficacy of tegavivint as a single agent in subjects with hepatocellular carcinoma as assessed by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)

OTHER OUTCOMES:
Evaluate efficacy of combination of tegavivint plus cabozantinib | Tumors will be assessed at baseline and every 8 weeks until end of treatment, an average of 1 year
  If sufficient clinical benefit is observed with tegavivint single agent, the efficacy of the combination of tegavivint plus cabozantinib will be evaluated using Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Evaluate efficacy of combination of tegavivint plus lenvatinib | Tumors will be assessed at baseline and every 8 weeks until end of treatment, an average of 1 year
  If sufficient clinical benefit is observed with tegavivint single agent, the efficacy of the combination of tegavivint plus lenvatinib will be evaluated using Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - City of Hope, Duarte, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Levine Cancer Institute, Charlotte, North Carolina
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- UHN - Princess Margaret Cancer Centre, Toronto, Ontario, Canada